CLINICAL TRIAL: NCT02053909
Title: Ticagrelor Antiplatelet Therapy to Reduce Graft Events and Thrombosis (TARGET Trial): Does Ticagrelor Improve Graft Patency After Coronary Bypass?
Brief Title: Ticagrelor Antiplatelet Therapy to Reduce Graft Events and Thrombosis
Acronym: TARGET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boca Raton Regional Hospital (Other)
Collaborators: AstraZeneca (Industry); Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Dr. Alexander Kulik, Cardiovascular Surgeon, Boca Raton Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Brilinta ISSBRIL0220
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Results first posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Saphenous Vein Graft Disease
Keywords: Saphenous vein graft disease; Coronary artery bypass graft surgery; Antiplatelet therapy; Coronary artery disease; Secondary prevention; Graft patency
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Active Comparator): One aspirin 81 mg capsule 2 times per day
  Interventions: Drug: Aspirin
- Ticagrelor (Active Comparator): One ticagrelor 90 mg capsule 2 times per day
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Aspirin
  Arms: Aspirin
Drug: Ticagrelor
  Other Names: Brillinta
  Arms: Ticagrelor

SUMMARY:
Saphenous vein graft disease remains an unresolved medical problem. Many vein grafts occlude in the first year after bypass surgery, leading to adverse cardiovascular outcomes, including recurrent angina, myocardial infarction, and the need for repeat coronary intervention. While aspirin is the standard antiplatelet treatment after CABG surgery, 10-20% of vein grafts continue to occlude despite contemporary secondary preventative therapy. Compared to aspirin and other antiplatelet therapies like clopidogrel, ticagrelor treatment leads to a more pronounced platelet inhibition, and may substantially improve graft patency following CABG compared to aspirin. No data has yet to be collected regarding the impact of ticagrelor on saphenous vein graft patency following CABG. In this context, the investigators seek to compare vein graft patency between patients randomized to receive aspirin therapy, the current standard of care, or ticagrelor treatment, starting in the early postoperative period, and continuing for 2 years after CABG.

DETAILED DESCRIPTION:
This clinical trial will be a randomized double-blind study focusing on ticagrelor antiplatelet therapy as a means of improving vein graft patency after CABG. Patients will be eligible if they have received at least 1 vein bypass graft at time of surgery. Patients will be randomized to receive either aspirin 81 mg bid or ticagrelor 90 mg bid. The aspirin and ticagrelor medications will be prepared in blinded capsules. Patients recovering from surgery will be eligible for study randomization within the first 5 postoperative days. Treatment will continue for 1 year, at which time patients will undergo a CT coronary angiogram to assess graft patency. Patients will then be invited to continue participating in the trial for 1 more year, and a repeat CT coronary angiogram will be performed at the 2 year postoperative time-point.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and/or male patients aged 18-90 years
3. Patients undergoing first-time CABG with at least 1 saphenous vein graft, irrespective of concurrent valve surgery

Exclusion Criteria:

1. Inability to provide informed consent
2. Pregnancy or seeking pregnancy
3. Patients undergoing redo-CABG
4. Serum creatinine >1.8 mg/dL (need for contrast with CT coronary angiogram)
5. Hypersensitivity or allergy to aspirin or ticagrelor
6. Anticipated need for postoperative anticoagulation with coumadin, dabigatran or rivaroxaban (mechanical valve, chronic atrial fibrillation, DVT/PE)
7. History of gastrointestinal hemorrhage
8. Active pathological bleeding
9. History of intracranial hemorrhage
10. Severe hepatic impairment
11. Current or anticipated use of strong CYP3A4 inhibitors (e.g. ketoconazole, clarithromycin, nefazadone, ritonavir, and atazanavir)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-09; Primary Completion 2020-08 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kulik, MD MPH, Principal Investigator — Boca Raton Regional Hospital
Locations (2):
- Boca Raton Regional Hospital, Boca Raton, Florida, United States
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Kulik A, Abreu AM, Boronat V, Kouchoukos NT, Ruel M. Impact of ticagrelor versus aspirin on graft patency after CABG: Rationale and design of the TARGET (ticagrelor antiplatelet therapy to reduce graft events and thrombosis) randomized controlled trial (NCT02053909). Contemp Clin Trials. 2018 May;68:45-51. doi: 10.1016/j.cct.2018.03.008. Epub 2018 Mar 15. PMID 29551675

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin: One aspirin 81 mg capsule 2 times per day
  Aspirin
- Ticagrelor: One ticagrelor 90 mg capsule 2 times per day
  Ticagrelor
Period: Overall Study
Arm/Group | Aspirin | Ticagrelor
Started | 123 | 127
Completed | 123 | 127
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aspirin: aspirin group
- Ticagrelor: ticagrelor group
- Total: Total of all reporting groups
Arm/Group | Aspirin | Ticagrelor | Total
Number analyzed (Participants) | 123 | 127 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (9.0) | 67.5 (9.3) | 68.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 23 | 39
  Male | 107 | 104 | 211
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Saphenous Vein Graft Occlusion
Description: The primary objective of this clinical trial will be to evaluate whether, as compared to usual aspirin treatment, ticagrelor early after CABG prevents saphenous vein graft occlusion 1 year after surgery, as assessed by computed tomography (CT) coronary angiography.
Time Frame: 1 year after surgery
Population: Vein graft occlusion reported as percentage
Measure: Number; unit: percentage of veins occluded
Units Other Than Participants: Vein grafts
Arm/Group | Aspirin | Ticagrelor
Number analyzed (Participants) | 123 | 127
Number analyzed (Vein grafts) | 172 | 166
percentage of veins occluded | 17.4 | 13.2

2. Secondary Outcome: Saphenous Vein Graft Stenosis
Description: The secondary objective of this clinical trial will be to evaluate whether, as compared to usual aspirin treatment, ticagrelor early after CABG prevents saphenous vein graft stenosis, defined as >50% narrowing of the graft, 1 year after surgery, as assessed by computed tomography (CT) coronary angiography.
Time Frame: 1 year after surgery
Population: Vein graft stenosis reported as percentage
Measure: Number; unit: percentage of veins stenosed
Units Other Than Participants: Vein grafts
Arm/Group | Aspirin | Ticagrelor
Number analyzed (Participants) | 123 | 127
Number analyzed (Vein grafts) | 172 | 166
percentage of veins stenosed | 4.1 | 4.2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Aspirin | Ticagrelor
All-Cause Mortality (participants affected / at risk) | 2/123 | 2/127
Serious Adverse Events (participants affected / at risk) | 5/123 | 9/127
Other Adverse Events (participants affected / at risk) | 0/123 | 0/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin (N=123) | Ticagrelor (N=127)
Bleeding (Blood and lymphatic system disorders) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT02053909/Prot_SAP_000.pdf